CLINICAL TRIAL: NCT00888303
Title: Randomized Controlled Trial on Efficacy of Preemptive 8 mg of Dexamethasone for Reducing Pain and Postoperative Nausea and Vomit After Thyroidectomy for Benign Disease.
Brief Title: Single Dose Steroid Before Thyroidectomy for Benign Disease to Improve Postoperative Nausea, Pain, and Vocal Function
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Misericordia e Dolce (Other)
Responsible Party: Principal Investigator, Marco Scatizzi, Md, Ospedale Misericordia e Dolce
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD123
Record Dates: First submitted 2009-04-23; First posted 2009-04-27 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomit; Postoperative Vocal Function; Thyroidectomy
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Vomiting | interventions — Dexamethasone; Saline Solution; Thyroidectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (dexamethasone) (Active Comparator): 20 minutes before total or partial thyroidectomy for benign disease a single dose of intravenous 8 mg/2mL of dexamethasone is administered
  Interventions: Drug: Dexamethasone; Procedure: Thyroidectomy, total or partial
- B (Control) (Placebo Comparator): 20 minutes before total or partial thyroidectomy for benign disease 100 mg of saline solutions are administered intravenous
  Interventions: Drug: saline solution; Procedure: Thyroidectomy, total or partial

INTERVENTIONS:
Drug: Dexamethasone — 20 minutes before total or partial thyroidectomy for benign disease a single dose of intravenous 8 mg/2mL of dexamethasone is administered
  Arms: A (dexamethasone)
Drug: saline solution — 20 minutes before total or partial thyroidectomy for benign disease 100 mg of saline solutions are administered intravenous
  Arms: B (Control)
Procedure: Thyroidectomy, total or partial — Surgical standard intervention

SUMMARY:
The purpose of this study is to evaluate the efficacy of 8 mg of dexamethasone administered prior surgery, to reduce pain, postoperative nausea and vomiting and to improve vocal function after thyroidectomy for benign disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients undergoing thyroidectomy

Exclusion Criteria:

* Patients who had received antiemetic therapy within 48 hours before surgery
* Patients with depression
* Chronic pain disorder
* Insulin-dependent diabetes mellitus
* History of severe and/or repeated PONV after previous minor surgery, that led to change from standard anesthetic protocol
* Pregnancy
* Age < 18 years
* Patients who had known malignant disease or had undergone previous thyroid or neck surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomit (PONV) measured in 4 grades | 8, 24, 32 and 48 hours after surgery

SECONDARY OUTCOMES:
Postoperative pain after thyroidectomy measured in a 0-100 Visual analog scale | 8, 24, 32 and 48 hours after surgery
Vocal function measured in a 0-100 Visual analog scale | 8, 24, 32 and 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marco Scatizzi, MD, Study Chair — Misericordia and Dolce Hospital; Marco Rettori, MD, Study Director — Misericordia and Dolce Hospital; Francesco Feroci, MD, Principal Investigator — Misericordia and Dolce Hospital
Locations (1):
- Misericordia and Dolce Hodpital, Prato, Po, Italy

REFERENCES:
- [Result] Worni M, Schudel HH, Seifert E, Inglin R, Hagemann M, Vorburger SA, Candinas D. Randomized controlled trial on single dose steroid before thyroidectomy for benign disease to improve postoperative nausea, pain, and vocal function. Ann Surg. 2008 Dec;248(6):1060-6. doi: 10.1097/SLA.0b013e31818c709a. PMID 19092351